CLINICAL TRIAL: NCT04707638
Title: Neurophysiological Characteristics of Subthalamic Deep-brain Stimulation (STN-DBS) Under General Anesthesia for Patients With Parkinson's Disease or Dystonia and Their Correlation With Prognosis
Brief Title: Neurophysiological Characteristics of Subthalamic Deep-brain Stimulation (STN-DBS)
Status: Withdrawn | Type: Observational
Why Stopped: Ethics application has not been completed yet
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: NS20201230
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease; Dystonia
Keywords: Parkinson Disease; Dystonia; deep brain stimultation; neurophysiological characteristics
MeSH Terms: conditions — Parkinson Disease; Dystonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease or dystonia patients: Patients with Parkinson's disease or dystonia and underwent STN DBS under general anesthesia in neurosurgery department
  Interventions: Other: No intervention used

INTERVENTIONS:
Other: No intervention used — No intervention used

SUMMARY:
The intraoperative neuroelectrophysiological signals were collected from patients undergoing STN-DBS under general anesthesia in the Neurosurgery Department of Wuhan union Hospital, and their preoperative conditions and postoperative efficacy will be evaluated.

DETAILED DESCRIPTION:
The intraoperative neuroelectrophysiological signals were collected from patients undergoing STN-DBS under general anesthesia in the Neurosurgery Department of Wuhan union Hospital, and their preoperative conditions and postoperative efficacy will be evaluated. The intraoperative neuroelectrophysiological signals would be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwentSTN-DBS in neurosurgery department of Wuhan Union Hospital.
2. Patients with Parkinson's disease or dystonia.

Exclusion Criteria:

1.Patients without enough follow-up length.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Parkinson's disease or dystonia and STN-DBS in neurosurgery department of Wuhan Union Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-11 (Estimated); Study Completion 2023-01-11 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | Two years postoperatively
  UPDRS has four parts: part I (nonmotor experiences of daily living, total score=16); part II (patient motor experience of daily living, total score=52); part III (clinician motor examination, total score=56); part IV (complications, total score=23). The total score of all the four parts is147. Higher scores means a worse outcome.
Burke Fahn Marsden's Dystonia Rating Scales(BFMDRS) | Two years postoperatively
  BFMDRS has two parts: BFMDRS movement part (BFMDRS-M) and BFMDRS disability part (BFMDRS-D). The total score of BFMDRS-M is 120 and the total score of BFMDRS-D is 30. Higher scores means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fu Peng, PHD, Principal Investigator — Neurosurgery department of Wuhan Union Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsai ST, Kuo CC, Chen TY, Chen SY. Neurophysiological comparisons of subthalamic deep-brain stimulation for Parkinson's disease between patients receiving general and local anesthesia. Tzu Chi Med J. 2016 Apr-Jun;28(2):63-67. doi: 10.1016/j.tcmj.2016.02.003. Epub 2016 Apr 10. PMID 28757724
- [Background] Yamada K, Goto S, Kuratsu J, Matsuzaki K, Tamura T, Nagahiro S, Murase N, Shimazu H, Kaji R. Stereotactic surgery for subthalamic nucleus stimulation under general anesthesia: a retrospective evaluation of Japanese patients with Parkinson's disease. Parkinsonism Relat Disord. 2007 Mar;13(2):101-7. doi: 10.1016/j.parkreldis.2006.07.008. Epub 2006 Oct 19. PMID 17055325